CLINICAL TRIAL: NCT05209737
Title: Trendelenburg As a First-line Intervention in Critically Ill, Sedated, Invasively Mechanically Ventilated, Hypotensive Patients: a Pilot Randomized Controlled Trial
Brief Title: Trendelenburg As a First-line Intervention in Critically Ill, Sedated, Invasively Mechanically Ventilated, Hypotensive Patients
Acronym: Trend
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Negovsky Reanimatology Research Institute (Other Government)
Responsible Party: Principal Investigator, Valery Likhvantsev, MD, Head of the Research V. Negovsky Reanimatology Research Institute, Negovsky Reanimatology Research Institute
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Trend
Record Dates: First submitted 2022-01-13; First posted 2022-01-27 (Actual); Last update posted 2024-11-14 (Actual); Status verified 2024-11

CONDITIONS: Hypotension; Shock
Keywords: Trendelenburg position; hypotension; hypovolemic shock; shock; head-down position
MeSH Terms: conditions — Hypotension; Shock | interventions — Head-Down Tilt

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Trendelenburg position (Experimental): Position: 10-degree Head-down position
  Interventions: Procedure: Trendelenburg position
- Semirecumbent position (Active Comparator): Position: 30-degree Head-up position
  Interventions: Procedure: Semirecumbent position

INTERVENTIONS:
Procedure: Trendelenburg position — A 10-degree head-down position will be used in this group
  Arms: Trendelenburg position
Procedure: Semirecumbent position — A 30-degree head-up position will be used in this group
  Arms: Semirecumbent position

SUMMARY:
A pilot randomized controlled trial to evaluate the efficacy and safety of Trendelenburg position in critically ill patients with hypotension, mainly patients with septic shock and post operative vasoplegia. The main aim is to assess whether Trendelenburg position can improve organ function through a reduction in the need of fluid infusion and dose of vasopressors.

Patients will be screened for participation in the study and eventually randomized based on a balanced randomization scheme (1:1) to Trendelenburg position up to 72 hours after intensive care unit (ICU) admission or Semirecumbent position (standard of care).

DETAILED DESCRIPTION:
Current consensus on circulatory shock management defines shock as a life-threatening, generalized form of acute circulatory failure associated with inadequate tissue perfusion. Recommended interventions to improve perfusion include early hemodynamic stabilization through fluid resuscitation, along with treatment of the cause of shock. If impaired cardiac function results in inadequate cardiac output and tissue hypoperfusion despite fluid therapy, vasopressor agents should be administered.

Nevertheless, fluid overload causes multi-organ edema, such as pulmonary edema or hepatic congestion. Moreover, the negative effects of fluid intravenous administrations were also studied on healthy volunteers during the years. Most of them showed the development of lung injury due to fluid administration.

In addition, vasopressors are also associated with poor outcomes. Described serious adverse effects include organ ischemia, tachyarrhythmias, and atrial fibrillation, leading to organ dysfunction and mortality.

The head-down position, also known as the Trendelenburg position, was originally used by the surgeon Friederich Trendelenburg to improve surgical exposure of pelvic organs. The Trendelenburg position became then a widely popular procedure in managing patients with hypotension and shock. The primary effect of the Trendelenburg position is an increase in cardiac output. Although the short term effect on blood pressure and CO is certain, there is no agreement on its benefit in terms of tissue perfusion and clinical outcome in critically ill hypotensive patients, as nobody has attempted the Trendelenburg position as first line management.

To date, the gold standard position for patients in ICU according to the latest ESICM guidelines to prevent ventilator-associated pneumonia is the semirecumbent position. Experts recommend elevating the head of the patient on the bed to a 20-45 degrees position, preferably >30 degrees position.

Critically ill patients with hypotension, mainly patients with septic shock and those with post-operative vasoplegia, may be a subgroup of patients, who would benefit from a head-down position if the risks of aspiration pneumonia are minimized. The Trendelenburg position might permit to avoid the deleterious side effects of fluids and vasoconstrictor administration.

The idea is that Trendelenburg position can improve organ function through a reduction in the need of fluid infusion and doses of vasopressors in hypovolemic, hypotensive ICU patients and therefore increase ventilator free days.

The main aim of this trial is to assess if Trendelenburg position can reduce time to severe hypotension resolution.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Admitted to the intensive care unit (ICU);
* Invasive mechanical ventilation;
* Pharmacological sedation;
* Mean arterial pressure (MAP)<65 mmHg or need of fluids infusion or any vasopressor in order to keep MAP > 65 mmHg
* Ongoing invasive and/or non-invasive arterial blood pressure monitoring
* Central venous line with central venous pressure (CVP) monitoring
* Naso-gastric tube in situ
* Indwelling bladder catheter
* Consent according to local ethical committee rules

Exclusion Criteria:

* Body mass index > 45
* Documented or suspected increased intracranial pressure, based on medical history or actual clinical condition (es. intracranial tumor, cerebral hemorrhage, encephalitis,...);
* Intra-abdominal hypertension >25 mmHg
* Documented or suspected increased intraocular pressure (any degree of glaucoma)
* Full stomach pyloric incontinence;
* Gastric stasis, defined as aspiration from the NG (nasogastric) tube of fecal, bloody, or green fluid greater than 100 mL upon insertion of the tube or within the preceding hour;
* Ongoing enteral nutrition
* No central line inserted or femoral central line only
* Not sutured known diaphragm lesions
* Known hiatus hernia
* Aortic bifurcation and/or lower extremity arterial stenosis ≥70% combined with stage 3 intermittent claudication (pain at rest)
* Patients who are not able to be investigated with a leg raising test (eg lower extremities fractures, backbone fractures or backbone pain or deformity, and those patients with large cannulas in the femoral vessels)
* Demand of specific postures (eg Trauma, fractures, backbone pain or deformity, patients with large cannulas in the femoral vessels, pronation including first pronation planned within 6 h…)
* Any device which, according to the clinician, makes it unfeasible or unsafe to put patients in the Trendelenburg position (eg Drainage in thoracic cavity)
* Mechanical Circulatory Support;
* (CHD) (Gleen, Fontaine);
* Advanced right ventricular dysfunction or advanced cardiac failure, in which volume overload worsens cardiac function (plateau stage in the Frank-Starling curve);
* Actual upper gastrointestinal bleeding
* Passive leg raising test non-responder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-01-31 (Actual); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-10-20 (Estimated)

PRIMARY OUTCOMES:
Time to severe hypotension resolution | 72 hours
  Time from randomization to timepoint in which MAP > 65 mmHg not requiring fluids or vasoactive drugs (VIS < 5), lasting > 1 hour, in the semirecumbent position

SECONDARY OUTCOMES:
Ventilator-free days at 28 days | 28 days
  28 days - number of days in which the mechanical lung ventilation was not used
ICU-free days at 28 days | 28 days
  28 days - number of days in which the patient was not in an intensive care unit
Restarting vasopressor/inotrope therapy | 28 days
  Using vasopressors and/or inotropes to maintain MAP ≥ 65 mm Hg after premature study termination (Vasoactive inotrope score > 5)
28-days mortality | 28 days
  all cause mortality
90-days mortality | 90 days
  all cause mortality
Acute kidney injury | 28 days
  number of patients who have acute kidney injury according to KDIGO classification
Acute liver failure | 28 days
  Rapid hepatic injury with coagulation derangements and hepatic encephalopathy and multi-organ failure in a patient with no history of liver disease
Ventilation-associated pneumonia | 28 days
  Pneumonia due to mechanical lung ventilation

CONTACTS AND LOCATIONS:
Locations (2):
- Russia (2):
  - Vishnevsky Center of Surgery, Moscow
  - Demikhov Municipal Clinical Hospital 68, Moscow

IPD SHARING:
Plan to Share IPD: No